CLINICAL TRIAL: NCT04417790
Title: Utility of Lung Ultrasound in the Estimation of Extravascular Lung Water in Pediatric Population- a Prospective Observational Study
Brief Title: Utility of Lung Ultrasound in the Estimation of Extravascular Lung Water in Pediatric Population
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr. Subhrashis Guha Niyogi, Fellow, Cardiac Anaesthesia, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: INT/IEC/2019/001513
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Pulmonary Congestion; Congenital Heart Disease; Post-Op Complication
Keywords: Lung ultrasound; Transpulmonary thermodilution
MeSH Terms: conditions — Heart Defects, Congenital; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Children under 12 years of age, Undergoing elective cardiac surgery for cyanotic or acyanotic congenital heart disease, Aristotle score ≤9, Giving prior written informed consent.
  Interventions: Diagnostic Test: Lung ultrasound and EVLW measurement by transpulmonary thermodilution.

INTERVENTIONS:
Diagnostic Test: Lung ultrasound and EVLW measurement by transpulmonary thermodilution. — Lung ultrasonography by 8 Quadrant protocol of Volpicelli et al. Transpulmonary thermodilution for extravascular lung water measurement

SUMMARY:
Increased extravascular lung water (EVLW) may increase mortality and morbidity in cardiopulmonary pathology. Many factors can cause increased extravascular lung water and pulmonary edema after cardiac surgery. This includes left ventricular failure, acute mitral regurgitation; systemic inflammatory response post-cardiopulmonary bypass, left to right shunts, transfusion associated acute lung injury, acute respiratory distress syndrome(ARDS) and sepsis.

The clinical assessment of lung water ranges from auscultation to radiological methods to invasive measurements like dye dilution or thermodilution studies.

Lung ultrasonography is the newest modality for noninvasive assessment of extravascular lung water. Lung ultrasound has been validated against auscultation, chest X-rays, CT chest as well as the bedside gold standard, transpulmonary thermodilution in adults.

Critically ill children are more susceptible to complications and worsened outcomes from increased EVLW.

Lung ultrasound correlates with clinical and radiological endpoints, but has not been validated against invasive objective measures like transpulmonary thermodilution.

Evaluation of transpulmonary thermodilution setups in the pediatric population has shown different normal values and cutoffs compared to adults, possibly due to differential rates growth and development.

It is aimed to investigate the correlation of Lung ultrasound based indices of extravascular lung water to invasive measures, assess optimum cutoffs to appropriate clinical endpoints and evaluate their sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* aged under 12 years,
* undergoing elective cardiac surgery for cyanotic or acyanotic congenital heart disease,
* Aristotle score ≤9,
* with prior written informed consent

Exclusion Criteria:

* Neonates,
* Children with any chest wall deformity,
* children with known lung disease, active infection,
* those weighing less than 3.5 kg.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cyanotic or acyanotic heart undergoing elective cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
correlation of lung USG B-line score with PICCO derived EVLW / EVLWI in pediatric cardiac surgical patients. | Till extubation or second post-operative day.
cutoffs for lung USG B-line score to Predict abnormal EVLWI values. | Till extubation or second post-operative day.

SECONDARY OUTCOMES:
trending ability of lung USG B-line score to predict PICCO derived EVLW / EVLWI in pediatric cardiac surgical patients. | Till extubation or second post-operative day.

CONTACTS AND LOCATIONS:
Overall Officials: Bhupesh Kumar, DM, Study Director — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education & Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided